CLINICAL TRIAL: NCT07174271
Title: Evaluation of Patient Satisfaction Following Anterior Composite Restorations: Immediate and One-Week Comparisons
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2023.816
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Composite Restorations
Keywords: composite restorations; Patient satisfaction; control sessions
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anterior Composite Restoration Group: Anterior Composite Restoration Group - Single cohort of healthy participants receiving direct anterior composite restorations on maxillary central/lateral incisors or canines. Eligibility included vital anterior teeth with healthy periodontium and an esthetic need (e.g., partial diastema closure or full-coverage/esthetic restoration) in 1-6 teeth. Procedures were performed under rubber-dam isolation with a standardized protocol in the same clinic. Patient-reported outcomes were collected immediately post-treatment and at 1-week using a patient-adapted, FDI-based questionnaire (A4, A3, A1, C15, C11; 0-10 scale).
  Interventions: Other: Patient satisfaction survey upon completion of anterior composite restorations and during follow-up sessions

INTERVENTIONS:
Other: Patient satisfaction survey upon completion of anterior composite restorations and during follow-up sessions — This study focuses on evaluating patient satisfaction with anterior composite restorations immediately after treatment and during subsequent follow-up visits. A structured questionnaire, based on modifications of the Fédération Dentaire Internationale (FDI) criteria, was administered to patients. Since the original FDI criteria were primarily designed for dentist-based evaluation, the questions were adapted into a patient-friendly format.
  Participants were asked to rate restorations across multiple domains, including esthetic anatomical form, color harmony and translucency, surface smoothness, the condition of the adjacent mucosa, and post-operative sensitivity and tooth vitality. Each parameter was scored on a numerical scale ranging from 0 to 10, allowing patients to express their subjective perception of treatment outcomes.
  By collecting these patient-reported outcomes both immediately after the procedure and during follow-up sessions, the study aims to provide a comprehensive under

SUMMARY:
Brief Summary

The goal of this observational study is to learn about patient-centered evaluations of anterior composite restorations performed under rubber dam isolation in adults treated at a university dental clinic. The main questions it aims to answer are:

How do patients rate their restorations immediately after treatment?

Do patient evaluations change one week after treatment compared to immediate assessment?

The study group consisted of vital maxillary central and lateral incisors and canines. Individuals requiring partial diastema or full-coverage restorations in one to six anterior teeth were included in the study. All restorative procedures were performed under rubber dam isolation in accordance with standard protocols. Restorations were immediately evaluated by patients after treatment and reassessed during a one-week follow-up session.

Evaluations were conducted using questions based on Fédération Dentaire Internationale (FDI) criteria. However, since the FDI criteria were primarily designed for dentists, it was not possible for patients to score the restorations according to the classic model. Instead, patient assessment was achieved by asking them to give a score between 0 and 10 for each category.

A total of 50 patients were included in the study, and the number of teeth evaluated varied depending on the number of anterior restorations performed on each patient.

In the questionnaire, patients were asked a total of five questions regarding the esthetic anatomical form , color harmony and translucency , surface smoothness, adjacent mucosal conditions , and post-operative sensitivity.

DETAILED DESCRIPTION:
In Marmara University Faculty of Dentistry Restorative Dentistry Clinic (hangi üniversite hangi klinik), a questionnaire was conducted. The study group vital maxillary central incisors, lateral incisors, and canines . The participants in the study comprised individuals who were in need of partial diastema or full-veneer restorations on one to six teeth in the anterior region. All restorative procedures were performed under rubber dam isolation in accordance with standard protocols. The restorations were evaluated by patients immediately following treatment and then re-evaluated during a one-week follow-up session. The restorations were evaluated by patients through questions prepared with reference to the FDI (Fédération Dentaire Internationale) Since the FDI criteria is designed for dental professionals, the patients were not able to score the restorations in a classical pattern. The patients scored the restorations giving a number from 0 to 10 for each category. In an effort to reduce variability and ensure standardisation, all restorative procedures were performed in the same clinical setting by a single experienced operator. In order to standardise lighting conditions, all evaluations were conducted at the same time of day and within the same clinical room. During the evaluation process, patients were provided with a large mirror, which facilitated a comprehensive assessment of their entire smile, as opposed to a small hand mirror that might not have allowed for such a thorough examination. The questionnaire study was started after the approval of the restoration completion by the department supervisors. Patients were not called for the questionnaire study outside of routine controls, evaluations were made immediately after the restorations are completed and at 1-week control sessions. The number of patients to be included in the study was determined by power analysis. A total of 50 patients are planned to be included in our study. The number of teeth to be evaluated will vary depending on the number of anterior restorations in total patients.

Inclusion criteria comprised patients aged 18 to 35 years with sufficient cognitive ability to comprehend and provide informed consent, clinically healthy gingiva and periodontium without bleeding or plaque accumulation, and vital maxillary incisors and canines free from clinical signs of irreversible pulpitis. Eligible participants presented with one to six teeth in the anterior maxillary region requiring either diastema closure or full veneer restorations, and all restorative procedures were performed under rubber dam isolation. Exclusion criteria included the presence of mental, cognitive, or physical disabilities; systemic diseases or serious medical risks such as cardiovascular disorders, diabetes mellitus, hypertension, or epilepsy; poor compliance or inability to maintain oral hygiene after treatment; and contraindications for rubber dam placement, including asthma, predominant mouth breathing, partially erupted or severely malposed teeth, or latex allergy. Patients with clinical or radiographic evidence of periapical pathology or pulpal pathology affecting either anterior or posterior teeth were also excluded.

In the questionnaire, a total of 5 questions were asked to the patients about esthetic anatomical form , color harmony and translucency, smoothness of the surface, adjacent mucosa, post-operative sensitivity and tooth vitality.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Sufficient cognitive ability to understand the consent process
* Clinically healthy gingiva and periodontium
* No bleeding or plaque accumulation
* Vital upper incisors and canines without signs of irreversible pulpitis (11-12-13-21-22-23)

Exclusion Criteria:

* Any disability (mental health conditions, mental disabilities and physical disabilities)
* Systemic diseases or serious medical risks (cardiovascular disorders, diabetes, hypertension, epilepsy)
* Compliance problems, inability to maintain hygiene after treatment
* Patients contraindicated for rubber dam placement (patient with asthma diagnosis, mouth breathing, partially erupted teeth, excessively malposed teeth and latex allergy)
* Signs of periapical pathology or pulpal posterior or anterior pathology

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of systemically healthy individuals aged 18 to 35 years who are capable of understanding and providing informed consent. Eligible participants must present with clinically healthy gingiva and periodontium, no bleeding or plaque accumulation, and vital maxillary incisors and canines (teeth 11, 12, 13, 21, 22, 23) without signs of irreversible pulpitis. Individuals with systemic diseases, disabilities, poor oral hygiene compliance, contraindications to rubber dam placement (e.g., asthma, mouth breathing, partially erupted or malposed teeth, latex allergy), or with signs of periapical or pulpal pathology will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Change in Patient Satisfaction Scores for Anterior Composite Restorations from Post-Treatment to 1-Week Follow-up | Immediately after treatment and at 1-week follow-up
  Patient satisfaction with anterior composite restorations was assessed immediately after treatment and at a 1-week follow-up visit. Evaluations were performed using a patient-adapted questionnaire based on the Fédération Dentaire Internationale (FDI) criteria. Because FDI criteria were originally designed for dentist-based assessment, the questions were simplified into a 0-10 numeric rating scale for patients.
  The questionnaire included five domains:
  Esthetic Anatomical Form Scale: 0-10(0 = very poor anatomical form, 10 = excellent anatomical form) Color Harmony and Translucency Scale: 0-10(0 = severe mismatch in color/translucency, 10 = perfect match with natural tooth) Surface Smoothnes Scale: 0-10(0 = very rough surface, 10 = perfectly smooth surface) Adjacent mucosal condition, Scale: 0-10(0 = severe inflammation, bleeding or pathology, 10 = healthy adjacent mucosa with no sign) Post-operative Sensitivity and Tooth Vitality Scale: 0-10 (0 = no sensitivity with preserved vitality)

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Istanbul Asya Kitasi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All data obtained without working will be shared if requested.
Supporting Information: Study Protocol